CLINICAL TRIAL: NCT03086707
Title: A Two-arm, Open Label, Prefatory Study to Explore Changes in Nasal Mucociliary Clearance Between Smokers and Never Smokers and to Standardize Nasal Scraping Procedure
Brief Title: Prefatory Study to Explore Changes in Nasal Mucociliary Clearance and to Standardize Nasal Scraping Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P1-CMS-01-US
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Smokers; Never Smokers
Keywords: nasal mucociliary clearance; saccharine transit time
MeSH Terms: interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cigarette smokers (Active Comparator): Subjects who have smoked at least 20 cigarettes per day for at least the past 5 years.
  Subjects will be allowed to use their own brand of non-menthol cigarettes. There will be no smoking restriction after the discharge at Visit 3 and during the 1 day follow-up period.
  Interventions: Other: Cigarette
- Never smokers (No Intervention): Subjects who have smoked less than 100 cigarettes throughout their lifetime and no cigarettes in the past 3 years.
  Subjects will not be allowed to smoke until discharge at Visit 3.

INTERVENTIONS:
Other: Cigarette — After enrollment, and between Visit 2 and Visit 3, the subjects will abstain from smoking for a period of 8 hours. At Visit 3, after the 8-hour smoking abstinence period, the subjects will smoke 1 single cigarette.
  Arms: Cigarette smokers

SUMMARY:
This study intends to evaluate the nasal mucociliary clearance (NMC) by determining the value obtained for saccharin transit time (STT) test over the course of 12 hours following a single cigarette use in adult smokers, to compare it relative to never smokers, and to examine the relationship between plasma nicotine levels and STT value in smokers and never smokers. Safety will also be monitored during the study.

The planned maximum study duration for a single study participant from Screening through completion of study will be 33 days.

ELIGIBILITY:
Inclusion Criteria to be met at Visit 1 and Visit 2:

* Male smokers aged ≥25 to ≤45 years old.
* Male never smokers aged ≥25 to ≤45 years old.
* Subject's BMI is comprised between 18.0 kg/m2 to 32.0 kg/m2, inclusive.
* Subject is healthy, as judged by the Investigator.

Additional Inclusion Criteria to allocate subjects in one of the two groups:

* Non-menthol cigarette smokers:

  * A positive urine cotinine test (≥200 ng/mL).
  * Smoked at least 20 cigarettes per day for at least the past 5 years.
  * eCO levels >10 parts per million (ppm).
  * No plans to quit smoking in the next 3 months.
* Never smokers:

  * Subject who has smoked less than 100 cigarettes throughout their lifetime and no cigarettes in the past 3 years.
  * A negative urine cotinine test (<200 ng/mL).
  * eCO levels ≤ 5 ppm.

Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Inability to taste sweet within 60 minutes in the STT test.
* Any condition the Principal Investigator or designee has cause to believe would interfere with the procedures for upper or lower airway function. This could include, but is not limited to, nasal/septum deviations, or nasal polyps or nasal allergies.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects will be enrolled.
Enrollment: 14 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Frank Lee, MD, Principal Investigator — Inflamax Research - Neptune
Locations (2):
- United States (2):
  - Inflamax Research - Neptune, Neptune City, New Jersey
  - Inflamax Research - Newark, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available.

REFERENCES:
- [Background] Schroeder A, Mueller O, Stocker S, Salowsky R, Leiber M, Gassmann M, Lightfoot S, Menzel W, Granzow M, Ragg T. The RIN: an RNA integrity number for assigning integrity values to RNA measurements. BMC Mol Biol. 2006 Jan 31;7:3. doi: 10.1186/1471-2199-7-3. PMID 16448564

RESULTS

PARTICIPANT FLOW:
Groups:
- Cigarette Smokers: Subjects who have smoked at least 20 cigarettes per day for at least the past 5 years.
  Subjects will be allowed to use their own brand of non-menthol cigarettes. There will be no smoking restriction after the discharge at Visit 3 and during the 1 day follow-up period.
  Cigarette: After enrollment, and between Visit 2 and Visit 3, the subjects will abstain from smoking for a period of 8 hours. At Visit 3, after the 8-hour smoking abstinence period, the subjects will smoke 1 single cigarette.
Period: Overall Study
Arm/Group | Cigarette Smokers | Never Smokers
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cigarette Smokers | Never Smokers | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (7.20) | 32.1 (4.30) | 33.0 (5.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.3 (7.18) | 85.9 (11.60) | 79.6 (11.35)

OUTCOME MEASURES:

1. Primary Outcome: Saccharin Transit Time at t0, Start of Product Use
Description: Before performing the test, each subject will spend approximately 15 minutes acclimatizing to the environment of the clinic. A 1-2 mm particle of saccharin will be placed under direct vision, approximately 1 cm behind the anterior end of the inferior turbinate. The position of the subject's head should be flexed approximately 10° by visual assessment.
  The saccharin transit time will be determined as the elapsed time in minutes and seconds from placement of the saccharin until the time the subject perceives a sweet taste.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
minutes | 8.4 [4.81 to 11.89] | 10.1 [4.05 to 16.21]

2. Primary Outcome: Saccharin Transit Time 4 Hours After Product Use
Description: as for outcome 1
Time Frame: Measured at 4 hours after product use.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
minutes | 8.0 [5.83 to 10.12] | 7.1 [1.98 to 12.28]

3. Primary Outcome: Saccharin Transit Time 8 Hours After Product Use
Description: as for outcome 1
Time Frame: Measured at 8 hours after product use.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
minutes | 9.9 [3.25 to 16.57] | 10.1 [3.03 to 17.11]

4. Primary Outcome: Saccharin Transit Time 12 Hours After Product Use
Description: as for outcome 1
Time Frame: Measured at 12 hours after product use.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
minutes | 8.6 [5.34 to 11.78] | 9.0 [2.61 to 15.47]

5. Primary Outcome: Concentration of Plasma Nicotine at t0, Start of Product Use
Description: Nicotine plasma concentrations will be measured using validated LC/MS/MS bioanalytical method.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
ng/mL | 18.8 [13.83 to 23.80] | 0.0 [0.00 to 0.00]

6. Primary Outcome: Concentration of Plasma Nicotine 4 Hours After Product Use
Description: Nicotine plasma concentrations will be measured using validated LC/MS/MS bioanalytical method.
Time Frame: Measured at 4 hours after product use.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
ng/mL | 4.6 [1.25 to 7.90] | 0.2 [NA to NA] — All subjects in the never smoker group presented a plasma value below the Lower Limit of Quantification at the study timepoints.

7. Primary Outcome: Concentration of Plasma Nicotine 8 Hours After Product Use
Description: Nicotine plasma concentrations will be measured using validated LC/MS/MS bioanalytical method.
Time Frame: Measured at 8 hours after product use.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
ng/mL | 2.8 [0.35 to 5.26] | 0.2 [NA to NA] — All subjects in the never smoker group presented a plasma value below the Lower Limit of Quantification at the study timepoints.

8. Primary Outcome: Concentration of Plasma Nicotine 12 Hours After Product Use
Description: The Nicotine plasma concentrations will be measured using validated LC/MS/MS bioanalytical method.
Time Frame: Measured at 12 hours after product use.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cigarette Smokers | Never Smokers
Number analyzed (Participants) | 7 | 7
ng/mL | 3.9 [-2.24 to 9.96] | 0.2 [NA to NA] — All subjects in the never smoker group presented a plasma value below the Lower Limit of Quantification at the study timepoints.

9. Secondary Outcome: Ribonucleic Acid Quantity (Right Nostril)
Description: Ribonucleic Acid quantity: concentration measured in the right nostril (RNA protect buffer) using two nasal scraping methods
Time Frame: Nasal scraping was performed at the final clinic visit, on Day 2, before checkout from the study.
Population: 10 study participants underwent nasal scraping using either method 1 or method 2.
Measure: Mean (Standard Deviation); unit: ng/uL
Groups:
- Nasal Scraping Method 1: Five study participants underwent nasal scraping using method 1.
- Nasal Scraping Method 2: Five study participants underwent nasal scraping using method 2.
Arm/Group | Nasal Scraping Method 1 | Nasal Scraping Method 2
Number analyzed (Participants) | 5 | 5
ng/uL | 47.5 (23.83) | 44.0 (43.77)

10. Secondary Outcome: Ribonucleic Acid Quantity (Left Nostril)
Description: Ribonucleic Acid quantity: concentration measured in the left nostril (Qiazol buffer) using two nasal scraping methods
Time Frame: Nasal scraping was performed at the final clinic visit, on Day 2, before checkout from the study.
Population: 10 study participants underwent nasal scraping using either method 1 or method 2.
Measure: Mean (Standard Deviation); unit: ng/uL
Arm/Group | Nasal Scraping Method 1 | Nasal Scraping Method 2
Number analyzed (Participants) | 5 | 5
ng/uL | 46.2 (36.64) | 57.9 (39.94)

11. Secondary Outcome: Ribonucleic Acid Quality (Right Nostril)
Description: Ribonucleic Acid quality assessed using the RNA integrity number: measured in the right nostril (RNA protect buffer) using two nasal scraping methods. RNA integrity Number is an algorithm for assessing RNA integrity and based on a numbering system from 1 to 10, with 1 being the most degraded profile and 10 being the most intact.
Time Frame: Nasal scraping was performed at the final clinic visit, on Day 2, before checkout from the study.
Population: 10 study participants underwent nasal scraping using either method 1 or method 2.
Measure: Mean (Standard Deviation); unit: RNA Integrity Number
Arm/Group | Nasal Scraping Method 1 | Nasal Scraping Method 2
Number analyzed (Participants) | 5 | 5
RNA Integrity Number | 8.6 (1.13) | 7.1 (1.91)

12. Secondary Outcome: Ribonucleic Acid Quality (Left Nostril)
Description: Ribonucleic Acid quality assessed using the RNA integrity number: measured in the left nostril (Qiazol buffer) using two nasal scraping methods. RNA integrity Number is an algorithm for assessing RNA integrity and based on a numbering system from 1 to 10, with 1 being the most degraded profile and 10 being the most intact.
Time Frame: Nasal scraping was performed at the final clinic visit, on Day 2, before checkout from the study.
Population: 10 study participants underwent nasal scraping using either method 1 or method 2.
Measure: Mean (Standard Deviation); unit: RNA Integrity Number
Arm/Group | Nasal Scraping Method 1 | Nasal Scraping Method 2
Number analyzed (Participants) | 5 | 5
RNA Integrity Number | 2.4 (0.54) | 2.3 (0.41)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the entire study duration of up to 7 months, with individual subject participation of a maximum of 33 days from the signature of the Informed Consent Form (ICF) until the end of the safety follow-up period.
Arm/Group | Cigarette Smokers | Never Smokers
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cigarette Smokers (N=7) | Never Smokers (N=7)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-05-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03086707/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/07/NCT03086707/SAP_001.pdf